CLINICAL TRIAL: NCT01449110
Title: A Randomized, 12 Months Follow-up, Dose-response, Placebo-Controlled, Double-Blind, 6-Arms Parallel Trial to Evaluate the Safety and Efficacy of a Resveratrol-enriched Grape Extract (Stilvid) in Primary and Secondary Patients of Cardiovascular Disease
Brief Title: Resveratrol-enriched Grape Extract (Stilvid) in Primary and Secondary Prevention of Cardiovascular Disease
Acronym: FUNGRAPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Collaborators: Hospital General Universitario Morales Meseguer (Other)
Responsible Party: Principal Investigator, Juan Carlos Espín de Gea, Research Professor, National Research Council, Spain
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CEBAS-CSIC-1
Record Dates: First submitted 2011-10-06; First posted 2011-10-07 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Cardiovascular Diseases
Keywords: Primary prevention; Secondary prevention; Resveratrol; Grape; Cardiovascular; Nutraceutical; Food complement
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Secondary Prevention; FcRA76 protein, Streptococcus sp. group A; whole grape extract; Primary Prevention; Ibc proteins, Streptococcus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo in PP (Placebo Comparator): Placebo arm in primary cardiovascular prevention (PP)
  Interventions: Dietary Supplement: Placebo in primary cardiovascular prevention (PP)
- Placebo in SP (Placebo Comparator): Placebo arm in secondary cardiovascular prevention (SP)
  Interventions: Dietary Supplement: Placebo in secondary prevention
- Grape extract in PP (Active Comparator): Grape extract obtained without resveratrol in primary cardiovascular prevention
  Interventions: Dietary Supplement: Grape extract in primary prevention (PP)
- Grape extract in SP (Active Comparator): Grape extract without resveratrol in secondary cardiovascular prevention
  Interventions: Dietary Supplement: Grape extract in SP
- Resveratrol-enriched grape extract in PP (Experimental): Resveratrol-enriched grape extract (Stilvid) in primary cardiovascular prevention
  Interventions: Dietary Supplement: Resveratrol-enriched grape extract in PP
- Resveratrol-enriched grape extract in SP (Experimental): Resveratrol-enriched grape extract (Stilvid) in secondary cardiovascular prevention
  Interventions: Dietary Supplement: Resveratrol-enriched grape extract in SP

INTERVENTIONS:
Dietary Supplement: Placebo in primary cardiovascular prevention (PP) — 12 months follow-up:
  1. capsule/day of placebo (350 mg maltodextrin) for 6 months
  2. capsules/day of placebo (350 mg + 350 mg maltodextrin) for 6 months
  Other Names: Group A-PP
  Arms: Placebo in PP
Dietary Supplement: Placebo in secondary prevention — 12 months follow-up:
  1. capsule/day (350 mg maltodextrin) for 6 months
  2. capsules/day (350 mg + 350 mg maltodextrin) for 6 months
  Other Names: Group A-SP
  Arms: Placebo in SP
Dietary Supplement: Grape extract in primary prevention (PP) — 12 months follow-up:
  1. capsule/day (350 mg grape extract) for 6 months
  2. capsules/day (350 mg + 350 mg grape extract) for 6 months
  Other Names: Group B-PP
  Arms: Grape extract in PP
Dietary Supplement: Grape extract in SP — 12 months follow-up:
  1. capsule/day (350 mg grape extract) for 6 months
  2. capsules/day (350 mg + 350 mg grape extract) for 6 months
  Other Names: Group B-SP
  Arms: Grape extract in SP
Dietary Supplement: Resveratrol-enriched grape extract in PP — Resveratrol-enriched grape extract (Stilvid) is obtained from grapes treated with UVC illumination. Similar polyphenolic content to conventional grape extract used in the arms 'Grape extract in PP' and 'Grape extract in SP' but containing 8 mg resveratrol.
  12 months follow-up:
  1. capsule/day (350 mg resveratrol-enriched grape extract) for 6 months
  2. capsules/day (350 mg + 350 mg resveratrol-enriched grape extract) for 6 months
  Other Names: Group C-PP; Stilvid is the key ingredient of Revidox (Actafarma, Spain)
  Arms: Resveratrol-enriched grape extract in PP
Dietary Supplement: Resveratrol-enriched grape extract in SP — Resveratrol-enriched grape extract (Stilvid) is obtained from grapes treated with UVC illumination. Similar polyphenolic content to conventional grape extract used in the arms 'Grape extract in PP' and 'Grape extract in SP' but containing 8 mg resveratrol.
  12 months follow-up:
  1. capsule/day (350 mg resveratrol-enriched grape extract) for 6 months
  2. capsules/day (350 mg + 350 mg resveratrol-enriched grape extract) for 6 months
  Other Names: Group C-SP; Stilvid is the key ingredient of Revidox (Actafarma, Spain)
  Arms: Resveratrol-enriched grape extract in SP

SUMMARY:
Resveratrol can exhibit benefits against cardiovascular diseases (CVDs) although the cardioprotective role of resveratrol as part of the human diet is not yet clear.

The aim of this trial is to evaluate the safety and efficacy of a resveratrol-enriched grape extract (Stilvid) in 150 patients from both primary and secondary cardiovascular prevention.

All the patients are gold-standard medicated (statins and others). A number of cardiovascular risk and safety markers will be evaluated after consuming 1 cap/day for 6 months and 2 caps/day for 6 additional months (total 12 months).

ELIGIBILITY:
Inclusion Criteria:

FOR PRIMARY PREVENTION:

* Lack of known cardiovascular disease (coronary acute syndrome, stable ischemic cardiopathy, peripheric arteriopathy and cerebrovascular diseases).
* Age between 18 and 80 years.
* The above criteria and diabetes mellitus or at least two of the following risk factors:

  1. Active smoking (10 cigarettes or more per day).
  2. Arterial hypertension (>= 140/90 mmHg).
  3. Hypercholesterolemia (LDL-cholesterol >130 mg/dL and/or HDL-cholesterol < 45 mg/dL in women and 50 mg/dL in men).
  4. Obesity (BMI > 30 kg/m2)

FOR SECONDARY PREVENTION:

* Stable patients who coronary syndrome, cerebrovascular accident or peripheric arteriopathy event occurred at least 6 months or more before the recruitment in the study. In addition:

  1. Age between 18 and 80 years.
  2. Ejection fraction of left ventricle >=45%.
  3. Functional status I or II according to the New York Heart Association.
  4. Clinic stability in the recruitment (no symptoms of thoracic pain during the last month).
  5. Lack of residual lesions without vascularization in those patients with catheterism.

     Exclusion Criteria:

     FOR PRIMARY AND SECONDARY PREVENTION:
* Patients who do not satisfy inclusion criteria and:

  1. Known allergy to grapes
  2. Pregnancy or lactation
  3. Intake of nutraceuticals

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-04; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Apolipoprotein-B | 6 months
oxidized LDL particles | 6 months
Plasminogen activator inhibitor type 1 (PAI-1) | 6 months and 12 months
Adiponectin | 6 months and 12 months

SECONDARY OUTCOMES:
C Reactive Protein | 6 months 12 months
Interleukin-6 | 6 months and 12 months
Interleukin-10 | 6 months and 12 months
Interleukin-18 | 6 months and 12 months
sICAM-1 | 6 months and 12 months
sVCAM-1 | 6 months and 12 months
D-dimer | 6 months and 12 months
Fibrinogen | 6 months and 12 months
Glycated hemoglobin | 6 months and 12 months
Glucose | 6 months and 12 months
GGT | 6 months and 12 months
AST | 6 months and 12 months
Urate | 6 months and 12 months
ALT | 6 months and 12 months
LDH | 6 months and 12 months
TSH | 6 months and 12 months
Thyroxine | 6 months and 12 months
ALP | 6 months and 12 months
CPK | 6 months and 12 months
Bilirubin | 6 months and 12 months
Creatinin | 6 months and 12 months
Albumin | 6 months and 12 months
Total cholesterol | 6 months and 12 months
LDL-cholesterol | 6 months and 12 months
HDL-cholesterol | 6 months and 12 months
Triglycerides | 6 months and 12 months
Hematocrit | 6 months and 12 months
Hemoglobin | 6 months and 12 months
Mean corpuscular volume | 6 months and 12 months
Leucocytes | 6 months and 12 months
Neutrophils | 6 months and 12 months
Lymphocytes | 6 months and 12 months
Eosinophils | 6 months and 12 months
Platelets | 6 months and 12 months
Mean platelet volume | 6 months and 12 months
Sedimentation rate volume | 6 months and 12 months
Gene expression profile in peripheral blood mononuclear cells (PBMNCs) | 6 months and 12 months
  Transcriptomic study. Evaluation of the gene expression profile in PBMNCs in a diabetic sub-group from Secondary prevention.
Total homocystein levels | 6 months and 12 months
  Total homocystein levels in plasma evaluated with UPLC-MS-QqQ
Measurement of atheroma plaque and carotid intim thickness | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Espín, PhD, Principal Investigator — National Research Council (CEBAS-CSIC, Murcia, Spain)
Locations (1):
- University Hospital Morales Meseguer, Murcia, Spain